CLINICAL TRIAL: NCT00369993
Title: A Randomised, Open Label, Five-way Crossover Study to Assess the Systemic Exposure of Fluticasone Propionate and Salmeterol From SERETIDE/ADVAIR 250HFA MDI Alone and With AeroChamber-Max Spacer and VOLUMATIC Both in Their Washed and Unwashed States in Adult Subjects With Mild or Intermittent Asthma
Brief Title: Spacer Comparison In Adult Asthmatics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SAS104449
Record Dates: First submitted 2006-08-28; First posted 2006-08-30 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: asthma; spacer
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol

SUMMARY:
Spacers are used by people with respiratory diseases who have problems using MDIs (metered dose inhalers). This study used fluticasone propionate/salmeterol to look at the pharmacokinetic profiles produced by different spacers in their washed and un-washed states.

DETAILED DESCRIPTION:
A randomised, open label, five-way crossover study to assess the systemic exposure of fluticasone propionate and salmeterol from SERETIDE™/ADVAIR™ 250 HFA MDI without spacer and with AeroChamber-Max spacer and VOLUMATIC™ both in their washed and unwashed states in adult subjects with mild or intermittent asthma.

ELIGIBILITY:
Inclusion criteria:

* Non-smoking with a BMI of 19 - 30
* Diagnosed with mild or intermittent asthma and taking medication for it.

Exclusion criteria:

* Taking oral corticosteroids or inhaled fluticasone propionate
* Have certain medical conditions or are not otherwise healthy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-03; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic profile of fluticasone propionate (in particular the area under the curve to time t and the maximum concentration)

SECONDARY OUTCOMES:
The pharmacokinetic profile of salmeterol and the time to maximum concentration of fluticasone propionate

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: SAS104449 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SAS104449 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SAS104449 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SAS104449 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SAS104449 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SAS104449 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SAS104449 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register